CLINICAL TRIAL: NCT02592733
Title: A Case Control Observational Study to Assess CYDAR Automated Overlay Guidance During EVAR
Acronym: CYDAR-IRAAA
Status: Completed | Type: Observational
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Tara Mastracci, Tara Mastracci, Clinical Lead, Aortic Surgery, Royal Free Hospital NHS Foundation Trust
Other Study IDs: IRAS171317
Record Dates: First submitted 2015-10-23; First posted 2015-10-30 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Historical Cohort: Patients who have undergone infrarenal endovascular repair at each centre in the past.
- Prospective Cohort: Patients undergoing infrarenal endovascular repair in the study using CYDAR in addition to the local angiography equipment.
  Interventions: Device: CYDAR

INTERVENTIONS:
Device: CYDAR — CYDAR is an automated image mask that is cloud based adn delivered to operating theatres over a secure network. It fuses preoperative images with intraoperative images to provide more accurate image guidance for the surgeon.
  Groups: Prospective Cohort

SUMMARY:
This is an observational trial to determine if use of fusion imaging in infrarenal endovascular aneurysm repair will decrease the radiation dose and improve patient safety for this procedure.

DETAILED DESCRIPTION:
The aorta is the main artery of the body. An aortic abdominal aneurysm (AAA) is defined as an abnormal dilatation of the aorta, based on a diameter of 3 cm or more, due to a weakness of the aortic wall that is prone to rupture, leading to a lifethreatening condition.

Once AAA diagnosed, a CTscan is required to assess the anatomy and if indicate an endovascular aneurysm repair (EVAR) is performed. This mini invasive procedure allows the exclusion of the AAA by positioning an endograft inside the aorta through a femoral access under live Xrays (fluoroscopy) guidance.

The Xrays are good at showing bones and radioopaque endovascular tools, but they do not show soft tissues like the aorta, and they produce flat (2D) images that superimpose all the 3D anatomical features. In order to see the aorta, physicians have to inject iodinated contrast during high quality imaging recording. One way to improve clinicians' perception of peroperative 3D vascular anatomy is to accurately overlay selected information from the preoperative CT scan (a 3D vascular mask) onto the live Xray image creating a '3D roadmap'. This advanced imaging application is currently available only in the latest expensive hybrid rooms. This trial will examine the clinical benefits of the first advanced imaging application allowing automated 3D overlay guidance during EVAR in any theatre. The software, combined with secure and certified cloud high performance computing, deduces the patient position from comparing the bony anatomy visible on the Xray to that on the patient's CT scan, enabling it to produce and update accurate and reliable overlays of the diagnostic CT 3D vascular mask throughout the operation (www.cydar.co.uk). Expected benefits include reducing the total Xray exposure of the patients and staff, reduced use of iodinated contrast (a major cause of kidney failure) and shortening procedure duration.

ELIGIBILITY:
Inclusion Criteria:

1. willing and able to give informed consent,and
2. aged 18 or older, and
3. been scheduled for endovascular repair of an infrarenal aortic aneurysm (EVAR), and
4. who have had a preoperative diagnostic CT scan, and
5. able (in the investigator's opinion) and willing to comply with the study requirements.

Exclusion Criteria:

1. Female participants who is pregnant or planning pregnancy during the course of the study.
2. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
3. Any patient requiring an associated procedure (iliac branch device implantation, renal or mesenteric angioplasty)
4. Ruptured AAA and emergency procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients deemed fit for infrarenal repair at one of 4 centres.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Radiation Dose (DAP) | This will be measured during the index operation. There will be no further radiation after that. Investigators expect that this study should take 12 months for full enrollment and analysis
  The Dose Area Product acquired in surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tara M Mastracci, MD, Principal Investigator — Royal Free Hospital NHS Foundation Trust

REFERENCES:
- [Derived] Maurel B, Martin-Gonzalez T, Chong D, Irwin A, Guimbretiere G, Davis M, Mastracci TM. A prospective observational trial of fusion imaging in infrarenal aneurysms. J Vasc Surg. 2018 Dec;68(6):1706-1713.e1. doi: 10.1016/j.jvs.2018.04.015. Epub 2018 May 24. PMID 29804734